CLINICAL TRIAL: NCT06881329
Title: Epigenome-wide DNA Methylation Profiling in Aneurysmal Subarachnoid Hemorrhage and Delayed Ischemic Neurologic Deficit
Status: Active, not recruiting | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Principal Investigator, Tomasz Klepinowski, Principal Investigator, Researcher at the Department of Neurosurgery, Pomeranian Medical University Szczecin
Other Study IDs: KB-0012/61/2021; 2021/41/N/NZ2/00844 (Other Grant/Funding Number: National Science Centre, Poland)
Record Dates: First submitted 2025-03-10; First posted 2025-03-18 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Delayed Cerebral Ischemia; Cerebral Vasospasm After Subarachnoid Hemorrhage; Intracranial Aneurysm
Keywords: aneurysmal subarachnoid hemorrhage; cerebral vasospasm; delayed ischemic neurologic deficit; delayed cerebral ischemia; aneurysm rupture; intracranial aneurysm
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm; Vasospasm, Intracranial; Aneurysm, Ruptured

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Subarachnoid hemorrhage with delayed ischemic neurologic deficit: This cohort includes patients diagnosed with aneurysmal subarachnoid hemorrhage who develop delayed ischemic neurologic deficit, defined as a new focal neurological deficit (paresis, dysphasia) or Glasgow Coma Scale decline of ≥2 points lasting >1 hour, not attributable to rebleeding, hydrocephalus, or hyponatremia. Diagnosis is confirmed with radiologic evidence of vasospasm on transcranial Doppler.
- Subarachnoid hemorrhage without delayed ischemic neurologic deficit: This cohort includes patients diagnosed with aneurysmal subarachnoid hemorrhage who do not develop delayed ischemic neurologic deficit. These patients exhibit no new focal neurological deficits and no Glasgow Coma Scale decline of ≥2 points beyond the acute phase of hemorrhage. Radiologic assessments confirm the absence of significant vasospasm on transcranial Doppler.
- Healthy controls without subarachnoid hemorrhage: This cohort consists of age-, sex-, race-, and ethnicity-matched healthy individuals with no history of aneurysmal subarachnoid hemorrhage (aSAH) or other neurological disorders. Participants were selected from a publicly available dataset (GSE246337).
  Blood DNA methylation profiles from this group serve as a baseline reference for comparison with aSAH patients

SUMMARY:
The goal of this observational study is to investigate DNA methylation changes in adults with bleeding from brain aneurysm, which is called aneurysmal subarachnoid hemorrhage (aSAH), and their association with delayed ischemic neurologic deficit (DIND). The main questions it aims to answer are:

Are there specific DNA methylation changes in peripheral blood that differentiate patients with aSAH from healthy individuals? Can DNA methylation changes in peripheral blood predict the development of DIND following aSAH? Researchers will compare blood DNA methylation profiles of aSAH patients to healthy controls and also do subgroup analysis of patients with DIND versus those without DIND to see if there are distinct methylation patterns associated with aSAH and DIND.

Participants with aSAH will:

* Have a blood sample collected shortly after admission to hospital.
* Undergo epigenome-wide DNA methylation profiling using the Infinium MethylationEPIC v2.0 BeadChip microarray.
* Be monitored for the development of DIND, defined by clinical symptoms and radiographic vasospasm.

This study aims to identify potential epigenetic biomarkers for aSAH susceptibility and DIND risk, which could improve early diagnosis and risk stratification in affected patients.

DETAILED DESCRIPTION:
This is a prospective observational case-control epigenome-wide association study (EWAS) designed to investigate DNA methylation changes in peripheral blood of patients with aneurysmal subarachnoid hemorrhage (aSAH) and their potential association with delayed ischemic neurologic deficit (DIND). The study aims to identify epigenetic biomarkers that may contribute to the pathophysiology of aSAH and DIND, as well as to assess whether these methylation patterns can serve as predictive markers for disease progression.

Study Design and Procedures

Population:

* Patients diagnosed with aSAH will be prospectively recruited from a tertiary neurosurgical center.
* The prospectively recruited patients will be anonymized and classified into DIND and non-DIND groups based on clinical and radiological criteria.
* Healthy control subjects will be matched for age, sex, race, and ethnicity using a publicly available dataset (GSE246337).

Data Collection and Processing:

* Peripheral whole blood samples (10 mL) will be collected within days 1-4 post-hemorrhage before the onset of vasospasm.
* DNA will be extracted using the salting-out method, followed by bisulfite conversion for methylation profiling.
* Genome-wide DNA methylation analysis will be performed using the Infinium MethylationEPIC v2.0 BeadChip microarray, covering ~850K CpG sites.
* Genotyping will be performed using Illumina Global Screening Array (GSA-24) v3.0 consisting of over 654 000 unique loci. PLINK v1.9 software will be used for the variant filtering and statistical analyses. We consider in this analysis only bi-allelic SNPs on autosomes. If this analysis yields significant associations between SNPs and DIND, methylation quantitative trait loci will be analyzed for examination of long-range interactions between relevant SNPs and differentially methylated CpG sites. These SNP-methylation interactions could provide unique and novel data on the vasospasm mechanism.
* Data processing will be performed using SeSAME R package with rigorous quality control measures, including:

  * Removal of probes spanning SNPs with a minor allele frequency >1%.
  * Filtering out probes with low bead count or detection p-values.
  * Exclusion of sex chromosome-associated probes and incorrectly mapped probes.

Diagnosis of DIND:

* DIND will be clinically defined as a new focal neurological deficit or Glasgow Coma Scale (GCS) decline of ≥2 points, lasting >1 hour and not attributable to other causes such as hydrocephalus, hyponatremia or rebleeding.
* Radiological confirmation of vasospasm will be based on cerebral angiography, CT angiography (CTA), or transcranial Doppler (TCD) findings.

Statistical Analysis Plan

Differentially Methylated Probes (DMPs):

* Identification of DMPs will be conducted using linear regression models, with Benjamini-Hochberg correction for multiple comparisons.
* Only CpG sites with an absolute Δβ-value >5% and an adjusted p-value <0.05 will be considered significant.
* Epigenetic clocks (Horvath clock, Hannum clock, SkinBlood clock, PhenoAge clock, GrimAge clock) will estimate biological age based on DNA methylation patterns at specific CpG sites

Machine Learning Analysis:

* LASSO regression will be applied for feature selection to identify methylation patterns most predictive of aSAH vs. healthy controls and DIND vs. non-DIND.
* Performance of the predictive models will be assessed using the R² metric.

Functional Enrichment Analysis:

* Gene Set Enrichment Analysis (GSEA) using "GENE2FUNC" function of Functional Mapping and Annotation of Genome-Wide Association Studies platform (FUMA GWAS) and Genomic Regions Enrichment of Annotations Tool (GREAT) will be used to identify biological pathways associated with significant methylation changes.
* Pathway analysis will focus on immune response, neuroinflammation, endothelial dysfunction, and phosphorous metabolism, as these processes have been implicated in aSAH pathophysiology.

Quality Assurance and Data Validation

Internal Data Validation:

* Automated data checks will be used to identify inconsistencies in methylation profiles.
* Comparative analysis against reference datasets will ensure that methylation patterns align with known biological mechanisms.

Source Data Verification:

* Methylation profiles will be cross-checked with publicly available databases to ensure consistency with previous epigenome-wide association studies.
* Patient demographic and clinical data will be verified against electronic medical records to ensure accuracy.

Handling Missing Data:

* If methylation data for specific CpG sites is missing or below detection thresholds, these sites will be excluded from analysis.
* Missing clinical data will be handled using multiple imputation methods to minimize bias.

Sample Size Justification

Cohort Composition:

* 61 aSAH patients (32 with DIND, 29 without DIND).
* 61 matched healthy controls from GSE246337.

The relatively small sample size was chosen based on previous EWAS studies in aSAH Limitations and Future Directions

Tissue-Specific Limitations:

o The study uses peripheral blood DNA, which may not fully reflect methylation changes in the cerebral vasculature. Future studies should validate findings in the arterial wall of the affected vessel using low-mortality rat models or cerebrospinal fluid.

DIND Subgroup Limitations:

o Due to the relatively small sample size, findings related to DIND will require external validation in larger cohorts.

Conclusion This study aims to provide novel insights into epigenetic changes associated with aSAH and DIND. By identifying differentially methylated CpG sites, the study seeks to improve biomarker discovery for early risk stratification and potential therapeutic targets in aSAH patients.

ELIGIBILITY:
Inclusion Criteria:

* subarachnoid hemorrhage in computed tomography (CT) scan
* ruptured aneurysm identified with angio-CT or digital subtraction angiography (DSA)
* aneurysm successfully embolized or clipped
* obtained informed consent
* Hunt-Hess grade ≤ 3 by day 14 (initial higher grade was allowed providing that patient improved to grade 3 or higher by day 14)

Exclusion Criteria:

* < 18 years old
* unable to sign informed consent
* diagnosis of idiopathic perimesencephalic subarachnoid hemorrhage
* aneurysm identified more than 14 days after the ictus
* more than 14 days at the Intensive Care Unit
* remaining in Hunt Hess grade 5 or World Federation of Neurological Surgeons (WFNS) grade 5 from admission up to post-bleeding day 14

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from a tertiary neurosurgical center at Pomeranian Medical University Hospital No. 1 in Szczecin, Poland. The study population includes consecutive adult patients diagnosed with aneurysmal subarachnoid hemorrhage who meet eligibility criteria. Patients are prospectively enrolled upon admission and followed for the development of delayed ischemic neurologic deficit.
  The control group consists of age-, sex-, race-, and ethnicity-matched healthy individuals selected from the publicly available GSE246337 dataset. This dataset serves as a reference population to identify epigenetic changes specific to aSAH.
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
DNA methylation changes associated with aneurysmal subarachnoid hemorrhage and delayed ischemic neurologic deficit | Within four days following the enrollment (as blood samples will be collected within days 1-4 post-hemorrhage). Methylation profiling and CpG analysis the entire batch will be conducted within one year following enrollment of the last participant
  Identification of differentially methylated CpG sites in peripheral blood DNA of patients with aneurysmal subarachnoid hemorrhage compared to healthy controls and to assess whether DNA methylation changes are associated with delayed ischemic neurologic deficit.
  The metrics and direction of DNA methylation changes will be reported as Δβ values

SECONDARY OUTCOMES:
Epigenetic clocks analysis and their association with chronological age in delayed ischemic neurologic deficit | Within four days following the enrollment (as blood samples will be collected within days 1-4 post-hemorrhage). Methylation profiling and epigenetic clock analysis will be conducted within one year following enrollment of the last participant
  Horvath clock, Hannum clock, SkinBlood clock, PhenoAge clock, GrimAge clock) will estimate biological age based on DNA methylation patterns at specific CpG sites. Pearson correlation of chronological age with the abovemention epigenetic clocks.

CONTACTS AND LOCATIONS:
Locations (1):
- Pomeranian Medical University Hospital No. 1, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
The study's epigenome-wide DNA methylation data from peripheral blood samples of aSAH patients and healthy controls will be shared via the Gene Expression Omnibus (GEO) repository. This dataset includes processed methylation profiles and metadata necessary for secondary analysis.
Supporting Information: Study Protocol
Time Frame: Data is already deposited in Gene Expression Omnibus repository (GSE290201) and will be available immediately upon publication. It will remain publicly accessible indefinitely according to GEO repository policies.
Access Criteria: The methylation dataset will be available for download from Gene Expression Omnibus (GEO) repository (GSE290201). Researchers will have an access to the data following GEO's standard data use agreements, which require appropriate citation of the original study.
URL: https://www.ncbi.nlm.nih.gov/geo/query/acc.cgi?acc=GSE290201

REFERENCES:
- [Derived] Klepinowski T, Przybylowicz P, Taryma-Lesniak O, Binkowski J, Lisman D, Ossowski A, Jarosz K, Sawicki M, Poncyljusz W, Taterra D, Latka K, Wojdacz TK, Sagan L. Epigenome-wide DNA methylation profiling in aneurysmal subarachnoid hemorrhage and delayed ischemic neurologic deficit: a prospective observational study. Int J Surg. 2026 Jan 1;112(1):832-843. doi: 10.1097/JS9.0000000000003324. Epub 2025 Sep 4. PMID 40905839
- Available data/document: Individual Participant Data Set: GSE290201 — https://www.ncbi.nlm.nih.gov/geo/query/acc.cgi?acc=GSE290201 — Gene Expression Omnibus repository